CLINICAL TRIAL: NCT01041040
Title: PETHEMA LAM07: Prospective, Multicenter, Uncontrolled Cohort Study to Analyze the Efficacy of a Risk Adapted Treatment Strategy, Including Gemtuzumab Ozogamicin (GO) During Consolidation, for Patients With Acute Myeloid Leukemia (AML)
Brief Title: LAM07: Study to Analyze the Efficacy of a Risk Adapted Treatment Strategy, Including Gemtuzumab Ozogamicin (GO) During Consolidation, for Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Josep Mª Ribera/Executive Secretary, PETHEMA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA-LAM07
Record Dates: First submitted 2009-12-28; First posted 2009-12-30 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Acute Myeloblastic Leukemia
Keywords: Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemtuzumab — gemtuzumab ozogamicin (GO) during consolidation for patients with acute myeloid leukemia (AML)

SUMMARY:
Prospective, multicenter, uncontrolled cohort study to analyze the efficacy of a risk adapted treatment strategy, including gemtuzumab ozogamicin (GO) during consolidation, for patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Patients will be stratified according to age in a first step, with a cut-point of 65 years old. For patients younger than 65 years old who achieve complete response, a second stratification will be made before first consolidation treatment. This second stratification will be performed according to the follow parameters: MDR at the end of induction, karyotype and molecular findings, including FLT3 internal tandem duplication (ITD) and NPM1 mutations. The following groups can be identified according to these parameters:

Group A:

Patients aged 65 or younger who are candidates for intensive chemotherapy.

Group A1:

Patients who are in first CR with negative MRD (less than 0.1%), good prognosis karyotype and, in the case of t(8;21) or inv(16), absence of mutations in the exon 17 of c-kit.

Group A2:

Patients who are in first CR with negative MRD (less than 0.1%), intermediate-risk karyotype, NPM1 positive and FLT3 negative.

Group A3:

Patients who are in first CR with negative MRD (less than 0.1%), intermediate-risk karyotype, absence of NPM1 mutations and who are negative for FLT3-ITD or FLT3-ITD positive with a ratio less than 0.8, regardless NPM1 status.

Group A4:

Patients who are in first CR with positive MRD (greater than 0.1%), t(8;21) or inv(16) with mutations in the exon 17 of c-kit, intermediate risk karyotype with positive FLT3-ITD and ratio greater or equal to 0.8 or high-risk karyotype.

Group B:

Patients over 65 years who are able to receive intensive chemotherapy.

TREATMENT SCHEDULE:

Treatment is tailored for each of the previously defined groups:

Group A:

Induction with Idarubicin and ARA-C in "3 +7" schedule (IDA 12 mg/m2 x 3 days and ARA-C 200 mg/m2 x 7 days).

Group A1:

Two consolidation cycles with ARA-C at a dose of 3 g/m2 on days 1, 3 and 5. Collection of peripheral blood stem cells (PBSC) after the first consolidation. Autologous stem cell transplantation (ASCT) with Busulphan 1 mg/kg/6 VO or 0,8 mg/kg/6 h IV (Busilvex®) from day -8 to -5; Etoposide 20 mg/kg/d from day -4 to -3 and ARA-C 3 g/m2/12 h from on days -3 and -2 (see criteria for HiDAC modification); and G-CSF 10 µg/kg/d from day -9 to -2 (BEA schedule). Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is not recommended in first CR in this group of patients.

Group A2:

First consolidation with Idarubicin and ARA-C at the same dose than induction plus GO 3 mg/m2 at day 1. Collection of PBSC after first consolidation. Second consolidation with ARA-C 3 g/m2 on days 1, 3 and 5 followed by ASCT with BEA conditioning. It is not recommended to perform Allo-HSCT, especially from alternative donors, in first CR.

Group A3:

First consolidation with Ida and ARA-C at the same dose than induction plus GO 3 mg/m2 at day 1. Collection of PBSC after first consolidation. Second consolidation with ARA-C 3 g/m2 on days 1, 3 and 5 followed by ASCT with BEA schedule if no HLA-identical sibling is available. Patients in this group are candidates for allo-HSCT in first CR if HLA-identical sibling is available. Allo-HSCT will be performed after first consolidation.

Group A4:

First consolidation with Ida and ARA-C at the same dose than induction plus GO 3 mg/m2 at day 1. Collection of PBSC after first consolidation. Second consolidation with ARA-C 3 g/m2 on days 1, 3 and 5 followed by ASCT with BEA schedule if no donor is available. Patients in this group are candidates for allo-HSCT in first CR, including alternative donors. Allo-HSCT will be performed after first consolidation or later if no donor is available at this time.

Group C:

Induction with Idarubicin and ARA-C "2 + 5" (IDA 12 mg/m2 x 2 days and ARA-C 200 mg/m2 x 5 days). Two consolidations with GO 3 mg/m2 day 1 and ARA-C 100 mg/m2 continuous infusion days 1 to 5.

AML CHARACTERIZATION AND SAMPLES COLLECTION:

To achieve a complete characterization of AML, inmunophenotype analysis (defining the pattern for MRD studies), cytogenetics, FISH for inv(16), t(8;21) and t(15;17), and molecular study for AML1/ETO, CBFβ/MYH11, NPM1 and FLT3-ITD will be performed in all cases. For FLT3-ITD, the ratio between the mutated and not mutated allele will be calculated.

During the phase of samples collection, DNA, RNA and viable cells will be stored.

ELIGIBILITY:
Inclusion Criteria:

For intensive chemotherapy:

1. Patients with the novo AML or secondary to MDS or previous treatment, regardless of age.
2. Signed written informed consent.
3. ECOG ≤ 2. If ECOG is greater than 2 due to AML, the patient can be included in the study.
4. LVEF > 40 % measured by means of echocardiography.
5. If background of respiratory disease (not related to the AML), risk factors or clinical criteria for COPD, the values of functional tests, including DLCO, should be greater than 50% of the expected.
6. Bilirubin, alkaline phosphatase and ALT < of 3 fold the upper normal value, providing that it is not due to the disease that motivates the treatment (AML).
7. Serum creatinine < 2,5 mg/dL providing that it is not due to the disease that motivates the treatment (AML).
8. In fertile aged women, negative pregnancy test and use of contraception methods are required.

Any patient who does not meet the inclusion and exclusion criteria for treatment with intensive chemotherapy can be evaluated individually when considering that could still obtain benefit from this treatment considering that could still obtain benefit from this treatment.

Criteria for GO administration in patient candidates for intensive chemotherapy

Same criteria for intensive chemotherapy, including the following specifications:

1. CD33 positive (more than 5 % of the leukemic population)
2. Exclusion for treatment with GO in cases of serious hepatic disease not due to AML.
3. In patients who are going to receive GO in two cycles, the second one will be only administrated if the toxicity due to the first cycle is recovered.
4. Though the GO administered dose is much lower than usual, it is recommended a period of two months between GO administration and hematopoietic stem cell transplantation (HSCT).

Criteria for the modification of high dose ARA-C

The dose of Ara-C in cycles containing HiDAC should be reduced in the following cases:

1. The hematopoietic recovery in the previous cycle has been longer than 28 days.
2. Presence in the previous cycles of a confluent maculopapular rash or drug-induced shedding.
3. More than 4 episodes of watery diarrhea per day.
4. Increase of 4 fold the previous normal value of aminotransferases or alkaline phosphatase in any of the cycles.
5. Total bilirubin greater than 3 mg/dL in any of the cycles.
6. Treatment with HiDAC will be definitively suspended (even that included in the BEA conditioning) when previous toxicity include severe cerebellar ataxia, confusion or another sign of central nervous toxicity that has not another clear explanation.

Exclusion Criteria:

1. Patients with blastic crisis of a chronic myeloid leukemia or other myeloproliferative syndromes evolving to acute leukemia.
2. Patients with AML in relapse.
3. Acute promyelocytic leukemia (M3 or M3v).
4. Absence of signed written informed consent.
5. ECOG ≥ 3 that it is not due to the disease that motivates the treatment (AML).
6. LVEF < 40 % determined by echocardiography study.
7. Values of respiratory functional tests, including DLCO, lower than 50% of the expected.
8. Bilirubin, alkaline phosphatase or GOT > 3 fold the upper normal value, providing that it is not due to the disease that motivates the treatment (AML).
9. Serum creatinine > of 2.5 mg/dL providing that it is not due to the disease that motivates the treatment (AML).
10. Positive pregnancy test or not use of effective contraception in fertile aged women.
11. Previous treatment with antileukemic chemotherapy, except hydroxyurea.
12. Presence of an active neoplasia different from the AML.
13. Presence of a serious psychiatric disease.
14. Positive HIV test.
15. Any other condition which limits or dissuades from the treatment with intensive chemotherapy, especially with anthracyclines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
To provide prognosis stratification of AML patients at the end of the induction treatment, based on minimal residual disease (MRD), cytogenetics and molecular findings.
To evaluate the efficacy and safety of a post-remission therapy strategy adapted to the prognosis of the patients, which optimizes the currently available treatment options and includes GO

SECONDARY OUTCOMES:
To analyze the different prognosis factors in AML, including the karyotype and the molecular findings at diagnosis and the MRD level at the end of the induction.

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel Angel, Dr, Study Chair — PETHEMA Foundation
Locations (1):
- Hoapital La Fe, Valencia, Valencia, Spain